CLINICAL TRIAL: NCT07035301
Title: A Study on the Safety and Feasibility of Using Low-dose Muscle Relaxants in Bronchoscopy Interventional Surgery
Brief Title: Application of Low-dose Muscle Relaxants in Bronchoscopic Interventional Procedures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harbin Medical University (Other)
Collaborators: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Shi xiaoqian, Graduate student, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ChiCTR2500098978
Record Dates: First submitted 2025-05-12; First posted 2025-06-25 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Disease of Respiratory System
Keywords: Interventional bronchoscopy; Airway control; Remimazolam; Remifentanil; Rocuronium
MeSH Terms: interventions — Saline Solution; Remifentanil; Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- normal saline (Placebo Comparator): During the induction of anesthesia, rocuronium is not used for anesthesia.
  Interventions: Drug: Normal Saline (Placebo); Drug: Lidocaine Intravenous Infusion; Drug: Remimazolam Tosilate; Drug: Remifentanil
- rocuronium bromide (Experimental): Using rocuronium for anesthesia during the induction phase of anesthesia.
  Interventions: Drug: Lidocaine Intravenous Infusion; Drug: Remimazolam Tosilate; Drug: Remifentanil; Drug: Rocuronium (0.15mg/kg/body mass)

INTERVENTIONS:
Drug: Normal Saline (Placebo) — During anesthesia induction, an equal volume of normal saline was used instead of rocuronium for anesthesia.
  Arms: normal saline
Drug: Lidocaine Intravenous Infusion — Lidocaine was administered at a dose of 0.5mg/kg for the induction of anesthesia.
Drug: Remimazolam Tosilate — Remimazolam was administered at a dose of 0.2 mg/kg for the induction of anesthesia.
Drug: Remifentanil — Remifentanil was administered at a dose of 3 micrograms per kilogram for the induction of anesthesia.
Drug: Rocuronium (0.15mg/kg/body mass) — Rocuronium was administered at a dose of 0.15mg/kg for the induction of anesthesia.
  Arms: rocuronium bromide

SUMMARY:
The purpose of this clinical trial is to observe the use of low-dose muscle relaxants in bronchoscopy intervention surgeries, compared with no muscle relaxants, in terms of the satisfaction of tracheal tube insertion after anesthesia induction, the incidence of laryngospasm, the grading of intraoperative cough and movement, and the recovery of patients after surgery. The main questions it aims to answer are:

* How safe and feasible is the use of low-dose muscle relaxants in bronchoscopy intervention surgeries?
* Is the muscle relaxant regimen better than the no-muscle-relaxant regimen?

Participants will:

* During anesthesia induction, the experimental group will use low-dose muscle relaxants for anesthesia, while the control group will not use muscle relaxants for anesthesia.
* Record the satisfaction of mask ventilation and the incidence of laryngospasm.

DETAILED DESCRIPTION:
Patients scheduled for elective bronchoscopy were randomly allocated to two groups: the muscle relaxant group and the non-muscle relaxant group.

Anesthesia Induction:

Muscle Relaxant Group: Intravenous injection of lidocaine (0.5 mg/kg), remimazolam (0.2 mg/kg), remifentanil (3 µg/kg), and rocuronium bromide (0.15 mg/kg).

Non-muscle Relaxant Group: Identical to the muscle relaxant group, except rocuronium bromide was replaced with an equivalent volume of normal saline.

In both groups, an appropriately sized laryngeal mask airway (LMA) was inserted using a standard technique.

Anesthesia Maintenance:

A continuous intravenous infusion of remimazolam was administered at a rate of 1 mg/kg/h, and remifentanil was infused at a rate of 0.25-0.5 µg/kg/min.

Primary Outcomes:The grading of chest wall rigidity, the incidence of difficult facemask ventilation, the incidence of SpO₂ < 92% during facemask ventilation, the incidence of laryngospasm, and the grading of cough and/or body movement during bronchoscope insertion.

Secondary Outcomes:Perioperative changes in blood pressure, heart rate, oxygen saturation, Bispectral Index (BIS), airway pressure, and end-tidal carbon dioxide (PETCO₂); LMA insertion conditions (time, number of attempts, and ease of insertion); dosage of anesthetic drugs used during the procedure; the incidence of intraoperative and postoperative adverse events; and the quality of postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective electronic bronchoscopic interventional surgery;
2. Age 18 years or older;
3. American Society of Anesthesiologists (ASA) I-III;
4. The duration of bronchoscopic surgery >=20min;
5. Through pre-anesthesia assessment, the patient/family member has informed consent and signed the consent form;
6. The general clinical information of the patient is complete.

Exclusion Criteria:

1. Patients with predictable difficult airway;
2. Small mouth opening (<2 transverse fingers);
3. Combined with severe cardiovascular disease, abnormal liver and kidney function;
4. Morbidly obese patients with body mass index (BMI) greater than 35kg/m^2;
5. Has a history of gastroesophageal reflux disease.
6. High risk of reflux aspiration;
7. Those who have a history of abnormal surgical anesthesia recovery in the past;
8. Patients with mental illness and previous allergies to conventional anesthetic drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
The incidence rate of laryngeal spasm | At the beginning of the operation
  Observe the degree of glottic opening (grade I: glottis opens well; grade II: glottis opens ≥⅔, mild laryngospasm; grade III: glottis opens ⅓-⅔, moderate laryngospasm; grade IV: glottis opens ≤⅓ or is completely closed, severe laryngospasm).Grades III and IV were defined as laryngospasm.
The incidence rate of choking cough when the bronchoscope first enters the trachea | At the beginning of the operation
  Grade 0: no choking cough response; grade 1: single mild choking cough response; grade 2: multiple mild choking cough responses(<=5s); grade 3: severe choking cough response(>5s).
Difficult facemask ventilation | During the process of anesthesia induction
  Grade A represented the presence of an end-tidal carbon dioxide (PETCO₂) waveform plateau; Grade B, the absence of a plateau but with a PETCO₂ value ≥ 10 mmHg; Grade C, the absence of a plateau and a PETCO₂ value < 10 mmHg; and Grade D, the absence of a detectable PETCO₂ waveform. Grades C and D were classified as difficult facemask ventilation.
Grading of chest wall rigidity | During the process of anesthesia induction
  Mild: No difficult ventilation but with stiffness of the limbs or abdominal wall.
  Moderate: Difficult ventilation accompanied by noticeable limb stiffness or abdominal wall rigidity.
  Severe: Inability to ventilate with significant limb stiffness or abdominal wall rigidity.
Grading of body movement during bronchoscope insertion | At the beginning of the operation
  Grade 1: Slight movement that does not interfere with the procedure.
  Grade 2: Pronounced movement that interferes with the procedure.
  Grade 3: Thrashing or vigorous movement that significantly interferes with the procedure.

SECONDARY OUTCOMES:
The severity of postoperative sore throat | When the patient regained consciousness (assessed up to 30 minutes after surgery)
  The patient's sore throat was evaluated using the visual analogue scale. A 10-cm movable ruler with 10 marks was used, with the two ends marked at 0 and 10 respectively. The patient was asked to mark the corresponding position on the ruler that represented their degree of pain. 0 represented no pain, and 10 represented extremely painful.
Dysphagia | When the patient regained consciousness (assessed up to 30 minutes after surgery)
  After the surgery, inquire whether the patient has any difficulty in swallowing.
Nausea | When the patient regained consciousness (assessed up to 30 minutes after surgery)
  After the surgery, ask the patient if they are experiencing nausea.
Number of laryngeal mask placements | During the process of anesthesia induction
  Record the number of times the laryngeal mask is inserted when it is placed.
Vomit | When the patient regained consciousness (assessed up to 30 minutes after surgery)
  After the surgery, ask the patient if they feel like vomiting.
Is it easy to insert the laryngeal mask? | During the process of anesthesia induction
  The difficulty level of inserting the laryngeal mask can be determined by observing the mouth opening during insertion, the resistance encountered during insertion, the presence or absence of choking and body movement, and the time taken for insertion. It is classified into four levels: simple, slightly difficult, difficult, and failed.
Bloating of stomach | When the patient regained consciousness (assessed up to 30 minutes after surgery)
  After the patient regains consciousness, ask the patient if they have any bloating in the stomach.
hoarseness | When the patient regained consciousness (assessed up to 30 minutes after surgery)
  After the patient regains consciousness, the presence of hoarseness in the patient is determined through communication with the patient.
Time of laryngeal mask placement | During the process of anesthesia induction
  The time required for laryngeal mask airway (LMA) insertion was measured from the initiation of the insertion attempt until correct placement was confirmed by the appearance of a normal end-tidal carbon dioxide (ETCO₂) waveform on capnography.
blood pressure | The time from when the patient enters the operating room until the patient finishes the surgery and leaves the operating room (up to 4 hours)
  Blood Pressure: The lateral pressure exerted by blood on the walls of blood vessels when it flows within them. Systolic blood pressure (SBP): The highest pressure in the arteries during the contraction of the heart (normal range: 90 - 120 mmHg). Diastolic blood pressure (DBP): The lowest pressure in the arteries during the relaxation of the heart (normal range: 60 - 80 mmHg).
heart rate | The time from when the patient enters the operating room until the patient finishes the surgery and leaves the operating room (up to 4 hours)
  Heart Rate: Number of heartbeats per minute (unit: beats per minute, bpm). . Normal resting heart rate: 60-100 beats per minute for adults.
  (For athletes or those who engage in long-term exercise, it can be as low as 40-50 beats per minute.)
oxyhemoglobin saturation | The time from when the patient enters the operating room until the patient finishes the surgery and leaves the operating room (up to 4 hours)
  Blood oxygen saturation (SpO2): The percentage of oxyhemoglobin (HbO2) in the blood relative to the total hemoglobin (Hb), reflecting the oxygenation status of the body. . Normal range: For healthy adults at rest, it is 95% - 100%. Anything below 90% indicates hypoxemia.
Bispectral index | The time from when the patient enters the operating room until the patient finishes the surgery and leaves the operating room (up to 4 hours)
  BIS is a method that analyzes the linear (frequency, power) and non-linear (phase, harmonic) components of electroencephalogram (EEG) data, converting them into quantitative indicators ranging from 0 to 100, which is used to assess the inhibitory or excitatory state of the cerebral cortex.
  Value range: 0 indicates no brainwave activity, and 100 represents a fully awake state.
  Core function: Primarily used for monitoring the depth of anesthesia, the level of sedation, and the state of consciousness, reducing the risk of intraoperative awareness.
airway peak pressure | The period from the start of anesthesia induction to the time when the patient leaves the operating room after the surgery is completed (up to 4 hours)
  Airway peak pressure is a very important parameter in mechanical ventilation, referring to the highest pressure value reached within one inhalation phase in the breathing circuit. The normal range is typically between 15 - 30 cmH2O. However, this varies depending on factors such as the patient's pathophysiological condition, ventilation mode, tidal volume, flow rate, and PEEP setting.
Airway platform pressure | The period from the start of anesthesia induction to the time when the patient leaves the operating room after the surgery is completed (up to 4 hours)
  Airway plateau pressure is a key parameter for evaluating the pressure that alveoli can withstand in mechanical ventilation, reflecting the pressure (plus the set PEEP) required to overcome the elastic resistance (compliance) of the lungs and chest cavity. It can more directly reflect the degree of alveolar expansion at the end of inspiration and predict the risk of ventilator-associated lung injury (such as pressure injury, volume injury). The generally accepted safe upper limit is ≤ 30 cmH₂O (including PEEP).
Carbon dioxide at the end of breathing | The period from the start of anesthesia induction to the time when the patient leaves the operating room after the surgery is completed (up to 4 hours)
  End-tidal carbon dioxide (EtCO₂) monitoring is a non-invasive, real-time, and continuous important technique. By measuring the partial pressure (usually expressed in mmHg or kPa) or concentration (%) of carbon dioxide in the exhaled gas of the patient, it reflects the ventilation function, metabolic status, and circulatory status. It is an indispensable monitoring method in anesthesia, intensive care, emergency rescue (especially cardiopulmonary resuscitation). Normal value: Adult: 35 - 45 mmHg (approximately 4.7 - 6.0 kPa).
Dosage of Anesthetic Drugs | Perioperative period
  The dosages of the following drugs were recorded throughout the perioperative period: lidocaine, remimazolam, remifentanil, rocuronium, propofol, ephedrine, norepinephrine, atropine, esmolol, ebrantil, dyphylline, and dexamethasone.
The satisfaction of the operating physician | 30 minutes after surgery
  The operating physician rated their satisfaction with the procedure on a scale from 1 to 10. The evaluation was based on procedural convenience, oxygenation stability (specifically, whether hypoxemia necessitated interruption of the procedure), and the overall smoothness of the workflow.
Anesthesiologist satisfaction | 30 minutes after surgery
  Anesthesiologist satisfaction with the procedure was rated on a scale from 1 to 10. The evaluation was based on the difficulty of airway management (particularly the frequency of interventions required to maintain adequate ventilation), the efficacy of oxygenation maintenance, and the incidence of adverse events.
Patient satisfaction | 30 minutes after surgery
  Patients rated their satisfaction with the procedure on a scale from 1 to 10. The rating was based on procedural comfort, the postoperative recovery experience, and their subjective perception of the sedation process.
Hypotension | Intraoperative
  The incidence of systolic blood pressure less than 80% of baseline.
Hypertension | Intraoperative
  The incidence of systolic blood pressure greater than 160 mmHg, exceeding 120% of baseline, or diastolic blood pressure greater than 100 mmHg.
Bradycardia | Intraoperative
  The incidence of heart rate less than 50 beats per minute (bpm).
Tachycardia | Intraoperative
  The incidence of heart rate greater than 100 beats per minute (bpm).
Severe cough | Intraoperative
  The incidence of cough grades 2 and 3.
Severe body movement | Intraoperative
  The incidence of body movement grades 2 and 3.
Airway rescue interventions | Intraoperative
  The frequency of the following airway rescue interventions was recorded: increasing the oxygen flow rate, performing manual ventilation, and administering an intravenous bolus of diprophylline (0.25 g).
Bronchospasm | Intraoperative
  The incidence of peak airway pressure greater than 30 cmH₂O.

CONTACTS AND LOCATIONS:
Overall Officials: SHI Jinghui SHI, Study Director
Locations (1):
- The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Yes
The original data sharing platform (IPD sharing platform) of ResMan, a clinical trial registration center of China, on June 30, 2028.
Supporting Information: Study Protocol, SAP, ICF, CSR
URL: http://www.medresman.org.cn/pub/cn/help.aspx